CLINICAL TRIAL: NCT03276338
Title: Using CBPR to Reduce HIV Risk Among Immigrant Latino MSM
Acronym: HOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00012292; 5R01MH087339-04 (NIH)
Record Dates: First submitted 2017-05-26; First posted 2017-09-08 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participation in the HOLA intervention designed to prevention HIV
  Interventions: Behavioral: HOLA
- Delayed-intervention (No Intervention): Delayed intervention with participation in HOLA intervention after follow-up data have been collected

INTERVENTIONS:
Behavioral: HOLA — To increase condom use and HIV testing
  Arms: Intervention

SUMMARY:
The intervention is based on social cognitive theory and theory of empowerment education and was developed using community-based participatory research (CBPR). This study is a result of a long-term community-university partnership that has used and will continue to use CBPR throughout all phases of research. A total of 21 Latino MSM in rural NC have been screened and recruited to serve as LHAs. The CBPR partnership selected LHAs based on qualities of natural helpers and informal leaders and having existing social networks of other Latino MSM. Eight members of each LHA's social network have been screened and recruited to participate as well. The LHAs, coupled with their social networks, have been randomized to intervention or delayed-intervention groups. LHAs (n=11) in the intervention group were trained and serve as LHAs within their social networks in Year 2. Delayed-intervention LHAs (n=10) receive the same LHA training and serve as LHAs within their social networks in Year 3. Quantitative assessment data is collected from each LHA (n=21) and the 8 members of his social network (n=189) longitudinally at: (1) baseline, (2) immediate post-intervention, and (3) 12-month follow-up. This is an "intent-to-treat" study, in which participant data are analyzed based on their randomization group.

The investigators hypothesize that participants in the HIV prevention intervention, relative to those in the delayed intervention comparison group, will demonstrate (1) increased self-reported use of condoms during sexual intercourse and (2) increased self-reported HIV testing.

The results and products from this study will be disseminated to inform public health practice, research, and policy. Results and products will include: (1) a Spanish-language intervention that is: culturally congruent and gender-specific; designed to reduce HIV risk among Latino MSM; and ready for dissemination and adaptation; (2) a deeper understanding of HIV risk and intervention among Latino MSM; and (3) insight into a CBPR process that includes community members, organizational representatives, and academic researchers.

DETAILED DESCRIPTION:
The goals of this study are to refine, implement, and evaluate a culturally relevant intervention designed to reduce the disproportionate HIV burden borne by Latino men who have sex with men (MSM) in the United States (US). This application is the culmination of ongoing research from an established partnership and was developed using community-based participatory research (CBPR). The proposed research refines an intervention that was developed, implemented, and evaluated using CBPR and was found effective in increasing condom use and HIV testing among heterosexual immigrant Latino men.1 Our CBPR partnership will refine the intervention based on findings from an R21 formative CBPR study among Latino MSM in rural North Carolina (NC) as well as ongoing insights provided by members of the partnership. CBPR will continue to be used to enhance the quality and validity of this research, continuing to equitably involve community members, organizational representatives, and academic researchers in all phases of the research. Together, the partners have developed the following specific aims for this proposal:

Aim 1: Refine a culturally relevant HIV prevention intervention designed to increase condom use and HIV testing among adult Latino MSM.

Aim 2: Implement and evaluate the effectiveness of the intervention by comparing Latino MSM in the intervention to those in the delayed-intervention comparison, using a study design recommended by members of the CBPR partnership.

The Specific Aims will be met by applying principles of CBPR to:

1. Refine the HoMBReS intervention, which has been found effective in increasing condom use and HIV testing among heterosexual Latino men, while retaining the integrity of intervention themes, concepts, and approaches;
2. Recruit and enroll adult male Latino lay health advisors (LHAs; total n=20) who represent 20 distinct social networks of Latino MSM within central NC;
3. Recruit and enroll 12 members from the social network of each of the 20 LHAs for a total of n=240 social network members;
4. Randomize the 20 LHAs, coupled with their social networks, into intervention and delayed-intervention comparison groups;
5. Train and support the LHAs in 2 waves (intervention and delayed-intervention) to serve as health advisors, opinion leaders, and community advocates;
6. Evaluate the impact of the intervention by comparing rates of change in condom use and HIV testing from baseline to immediate post-intervention between those in the intervention group (10 LHAs; 120 social network members) and their peers in the delayed-intervention group (10 LHAs; 120 social network members), who will not have been exposed to the intervention, using an interviewer-administered assessment;
7. Evaluate the sustainability of intervention by comparing rates of change in condom use and HIV testing from immediate post-intervention to a 12-month follow-up using data from both the intervention and delayed-intervention groups who will all have been exposed to the intervention; and
8. Interpret and disseminate findings to community members, other key stakeholders, and policy leaders at the local, regional, and national levels.

This study will advance the field of HIV prevention research by refining, implementing, and evaluating an intervention for Latino MSM, who are disproportionately affected by HIV. Currently, there are few HIV prevention interventions with evidence of efficacy and none tailored to the unique and growing Latino immigrant communities currently settling in the southeastern US. Moreover, although LHA interventions are widely promoted, outcome data supporting LHA interventions as an approach to health promotion and disease prevention are limited. Our HoMBReS intervention, which was developed, implemented, and evaluated using CBPR, uses an LHA approach and has evidence of effectiveness.1 The investigators propose to refine it to fill important gaps in both the science and the practice of HIV prevention. The results and products from this study will be disseminated to inform public health practice, research, and policy. Results and products will include: (1) a Spanish-language intervention that is: culturally relevant and gender-specific; designed to reduce HIV risk among Latino MSM; and ready for dissemination and adaptation; (2) a deeper understanding of HIV risk and prevention among Latino MSM; and (3) insight into a research process that includes community members, organizational representatives, and academic researchers.

Study hypotheses. The investigators hypothesize that compared to participants in the delayed-intervention group, participants in the intervention group will demonstrate (a) increased self-reported use of condoms during sexual intercourse; and (b) increased self-reported HIV testing. The investigators also hypothesize that the sustainability of intervention will continue through 12-month follow-up (24 months after the Navegantes are trained).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Latino or Hispanic;
* be 18 years of age;
* report MSM behavior since age 18;
* have some Spanish-language literacy;
* and provide informed consent.

To be eligible to participate as a social network member of a Navegante, a participant must:

* self-identify as Latino or Hispanic;
* be 18 years of age;
* report MSM behavior since age 18;
* and provide informed consent.

Exclusion Criteria:

* having participated in the HoMBReS or HoMBReS-2 interventions, or in the refinement of the HOLA intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender identity is an inclusion criterion
Enrollment: 186 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Change in condom use | 4 months
  Evaluate the amount of condom use at from baseline to 4 months.

SECONDARY OUTCOMES:
Change in HIV status | 12 months
  Evaluate the change in HIV status from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rhodes, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided